CLINICAL TRIAL: NCT01592682
Title: "Creating Smokefree Living Together": Smokefree Counseling Intervention for Chinese Smokers and Household Nonsmokers
Brief Title: Creating Smokefree Living Together for Chinese Household Pairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 261778; RSGT-10-114-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2012-04-26; First posted 2012-05-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Smoking; Smoke Exposure
Keywords: tobacco; secondhand smoke; Chinese; NNAL
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Household pairs that are assessment only and receive usual care of local in-language smoking cessation resource referral including quitline.
- Smokefree counseling (Experimental): Household pairs assigned to smokefree counseling intervention, consisting of group education sessions, tobacco exposure lab report, individual follow-up phone calls.
  Interventions: Behavioral: Smokefree counseling

INTERVENTIONS:
Behavioral: Smokefree counseling — Smokefree counseling intervention involves group education sessions, follow-up phone calls, tobacco exposure lab report. Comparison is usual care with referral to local in-language smoking cessation services including quitline.
  Arms: Smokefree counseling

SUMMARY:
This is a trial of household pairs of a Chinese smoker and nonsmoker randomized either to a smoke-free educational intervention or self-help control group. The smokefree educational intervention includes group education about smokefree environments and smoking cessation, follow-up phone calls, and tobacco exposure lab reports. The control group is referred to usual care with local in-language smoking cessation classes or quitline, and is otherwise assessment only. The investigators hypothesize that pairs in the intervention group will have higher rates of tobacco cessation and elimination of smoke exposure, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Chinese Americans who primarily speak Chinese
* Self-identified current smoker men and nonsmoker women
* Pair lives in same household

Exclusion Criteria:

* Current smoker women
* Nonsmoker men

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 12 months
Elimination of secondhand smoke exposure | 12 months
  Nonsmoker
Urine NNAL (4-(Methylnitrosamine)-1-(3-pyridyl)-1-butanol) | 12 months
  Smoker and nonsmoker; NNAL is a tobacco-specific carcinogen

SECONDARY OUTCOMES:
Cigarette consumption | 12 months
  Smoker
Rule for no smoking in home | 12 months
  Smoker and nonsmoker
Reduction in secondhand smoke exposure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisa K Tong, MD, MA, Principal Investigator — University of California, Davis
Locations (1):
- Chinatown Public Health Center, San Francisco, California, United States

REFERENCES:
- [Derived] Chang E, Dove M, Saw A, Tsoh JY, Fung LC, Tong EK. Home Smoking Bans and Urinary NNAL Levels to Measure Tobacco Smoke Exposure in Chinese American Household Pairs. Int J Environ Res Public Health. 2021 Jul 20;18(14):7682. doi: 10.3390/ijerph18147682. PMID 34300133